CLINICAL TRIAL: NCT01895049
Title: Comparison Between Two Tacrolimus-based Immunosuppressant Regimens and Induction With Thymoglobulin in Kidney Transplants From Deceased Donors With Expanded Criteria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helio Tedesco Silva Junior (Other)
Collaborators: Novartis (Industry); Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Helio Tedesco Silva Junior, PhD, Hospital do Rim e Hipertensão
Organization: Hospital do Rim e Hipertensão (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ABR32T
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Kidney Transplantation; Cytomegalovirus
Keywords: Tacrolimus; Everolimus; Cytomegalovirus; Thymoglobulin; Deceased donors; Expanded criteria
MeSH Terms: interventions — Neoadjuvant Therapy; thymoglobulin; Prednisone; Everolimus; Mycophenolic Acid

ARMS (2):
- Mycophenolate sodium (Active Comparator): Induction therapy with Thymoglobulin, prednisone, mycophenolate sodium, and late introduction of tacrolimus
  Interventions: Drug: Induction therapy with Thymoglobulin, prednisone, mycophenolate sodium and late introduction of tacrolimus
- Everolimus (Experimental): Induction therapy with Thymoglobulin, prednisone, everolimus, and late introduction of tacrolimus.
  Interventions: Drug: Induction therapy with Thymoglobulin, prednisone, everolimus and late introduction of tacrolimus

INTERVENTIONS:
Drug: Induction therapy with Thymoglobulin, prednisone, everolimus and late introduction of tacrolimus
  Arms: Everolimus
Drug: Induction therapy with Thymoglobulin, prednisone, mycophenolate sodium and late introduction of tacrolimus
  Arms: Mycophenolate sodium

SUMMARY:
The disparity between supply and demand for organs has stimulated the development of strategies to increase the availability of kidney grafts. Such strategy involves the use of kidneys with expanded donor criteria (EDC). This is a study initiated by the investigator, open, prospective, randomized, single center designed to compare the safety and efficacy of two immunosuppressive regimens based on thymoglobulin, tacrolimus and everolimus versus thymoglobulin, tacrolimus and mycophenolate sodium in renal transplant recipients with donor criteria expanded.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years) candidates to renal transplant with expanded criteria deceased donors;
* Low risk of acute rejection, defined as first kidney transplant recipients and Panel Reactive Antibody (PRA) <50%.
* Signature of the informed consent form (ICF)

Exclusion Criteria:

* Patients receiving immunosuppressive therapy before transplantation;
* Patients who have received an investigational drug within last 30 days;
* Patients with a known contraindication to the administration of an anti-thymocyte globulin;
* Patients with a positive test for human immunodeficiency virus (HIV);
* Patients who had cancer (except non-melanoma skin cancer) within last two years;
* Pregnant women, breastfeeding women, and women of childbearing potential unwilling to use condoms or oral contraceptives will be excluded;
* Patients with any Panel Reactive Antibody (PRA) equal to or higher than 50%, class I or class II, will also be excluded;
* Patients with positive test for parasites (protozoa and helminths).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
Incidence of CMV disease | 1 year
  Incidence of CMV disease or infection during the first year of transplantation.

SECONDARY OUTCOMES:
incidence of treatment failure | 1 year
  To compare the two immunosuppressive regimens for the incidence of treatment failure defined as the composite endpoint of BPAR (biopsy-proven acute rejection), graft loss, death and loss to follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital do Rim e Hipertensao, São Paulo, Brazil

REFERENCES:
- [Derived] Oliveras L, Lopez-Vargas P, Melilli E, Codina S, Royuela A, Coloma Lopez A, Fava A, Manonelles A, Couceiro C, Lloberas N, Cruzado JM, Montero N. Delayed initiation or reduced initial dose of calcineurin-inhibitors for kidney transplant recipients at high risk of delayed graft function. Cochrane Database Syst Rev. 2025 Apr 8;4(4):CD014855. doi: 10.1002/14651858.CD014855.pub2. PMID 40197799
- [Derived] Ferreira AN, Felipe CR, Cristelli M, Viana L, Mansur J, de Paula M, Wagner D, de Marco R, Gerbase-DeLima M, Proenca H, Aguiar W, Medina-Pestana J, Tedesco-Silva Junior H. Prospective randomized study comparing everolimus and mycophenolate sodium in de novo kidney transplant recipients from expanded criteria deceased donor. Transpl Int. 2019 Nov;32(11):1127-1143. doi: 10.1111/tri.13478. Epub 2019 Aug 27. PMID 31278785